CLINICAL TRIAL: NCT00302731
Title: Prospective Double Blind Evaluation of Bioidentical Hormones
Brief Title: Bioidentical 'Natural' Hormone Evaluation in Early Menopause
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Jeanne Drisko, MD, CNS, FACN (Other)
Collaborators: Private Foundation through KU Endowment (Unknown); University of Kansas (Other)
Responsible Party: Sponsor-Investigator, Jeanne Drisko, MD, CNS, FACN, Director Integrative Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9941
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Menopause
MeSH Terms: interventions — Estradiol; Estriol; Progesterone; Estrogens, Conjugated (USP); Medroxyprogesterone Acetate; Prempro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1 equine estrogens m-progesteroneacetate (Active Comparator): Menopausal women in first seven years of menopause randomized to arm 1 receive conjugated equine estrogens 0.45 mg combined with medroxyprogesteroneacetate 1.5 mg placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
  Interventions: Drug: equine estrogens m-progesteroneacetate
- 2 estradiol estriol progesterone (Experimental): Menopausal women in first seven years of menopause randomized to arm 2 estradiol .5mg, estriol 2.0mg, progesterone 100mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
  Interventions: Drug: Estradiol , estriol , progesterone
- 4 estradiol progesterone (Experimental): Menopausal women in first seven years of menopause randomized to arm 4 estradiol 0.5 mg, progesterone 100 mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
  Interventions: Drug: estradiol, progesterone
- 3 estriol progesterone (Experimental): Menopausal women in first seven years of menopause randomized to arm 3 estriol 2.5mg, progesterone 100mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
  Interventions: Drug: estriol, progesterone

INTERVENTIONS:
Drug: Estradiol , estriol , progesterone
  Other Names: compounded bioidentical hormone
  Arms: 2 estradiol estriol progesterone
Drug: estradiol, progesterone
  Other Names: compunded bioidentical hormone
  Arms: 4 estradiol progesterone
Drug: estriol, progesterone
  Other Names: compounded bioidentical hormone
  Arms: 3 estriol progesterone
Drug: equine estrogens m-progesteroneacetate
  Other Names: Premarin and Provera; Prempro
  Arms: 1 equine estrogens m-progesteroneacetate

SUMMARY:
Prospective double blind pilot study comparing bioidentical 'natural' hormones to low-dose PremPro. Forty participants will be enrolled. The purpose of this study is to try to gather early information about safety when "natural" or bioidentical hormones are used during early menopause.

DETAILED DESCRIPTION:
In spite of warnings regarding safety and adverse events widely publicized after the Women's Health Initiative (WHI), women continue to seek hormone replacement therapy for a variety of reasons. Increased cardiovascular events identified in WHI are an important concern for considering menopausal hormone replacement. There is the belief the 'natural' or bioidentical hormone replacement therapy could provide a safe alternative to widely used synthetic hormone replacement therapy. However, this has never been studied with any rigor and health care providers can not adequately advise patients seeking 'natural' bioidentical hormone therapy.

This feasibility pilot study is designed as a prospective double blind study comparing 4 groups of women who are within 7 years of menopause. There will be 10 women in each of the 4 groups with a total of 40 women enrolled and these women will be treated for 12 months.

The Long-Term Goal is to provide health care practitioners and consumers with evidence-based recommendations for the use of bioidentical hormone replacement. The Short-Term Goal of this pilot study is to determine if it is feasible to conduct a study in bioidentical hormones and obtain information that could lead to a larger more definitive study. We would like to provide safety information for bioidentical hormone use by evaluating surrogate markers for cardiovascular disease (lipid levels), with secondary evaluation of breast (mammogram) and uterus (endovaginal ultrasound), and to collect information about bone preservation.

The information gained from this trial will provide information for a future trial to test the hypothesis that bioidentical hormone replacement therapy provides a safe alternative to standard hormone replacement therapy: To determine if bioidentical hormone replacement therapy is associated with improved lipid profiles (surrogate marker for cardiovascular disease) when compared to Prempro. This will be determined by evaluating lipid levels at baseline and during the 12-month treatment period.

Secondary hypotheses will also be evaluated in the future to include:

1. To determine if bioidentical hormone replacement therapy provides improved short-term risk profiles for uterine and breast health when compared to Prempro. This will be accomplished by requiring mammograms and endovaginal ultrasounds at baseline and the end of the 12-month treatment period.
2. To determine if there is bone loss when using bioidentical hormone replacement when compared to Prempro. This aim will be evaluated by Dexa bone scan at baseline and at 12 months.

Subjects will randomly be assigned to one of the four arms of the study for the 12 months of treatment. The standard of care arm will consist of 10 women receiving in a double blind fashion low-dose Prempro. There will be 3 treatment arms consisting of different combinations of E2 estradiol and/or E3 estriol, all combined with bioidentical progesterone. These 3 arms will each have 10 subjects randomized and the bioidentical hormone delivered in a double blind fashion. Since the gold standard for treatment is the conventional arm (Prempro), we will compare each bioidentical arms to the gold standard. This comparison will occur at the end of 12 months of treatment. In this pilot study, we also wish to collect preliminary data about the comparisons between the 3 bioidentical hormone arm and the conventional arm. This is necessary because there is currently anecdotal evidence that E3 alone without combination with E2 may constitute adequate therapy in spite of its low biological activity at the estrogen receptor. The use of high doses of E3 with or without E2 is in common use by complementary and alternative practitioners.

It is expected in this small pilot study that bioidentical hormone will provide an adequate short-term safety profile for cardiovascular, breast and uterine health that will provide guidance for a larger trial that is longer in duration. It is also expected that bone density may be maintained by bioidentical hormone replacement when compared to Prempro. There may not be sufficient numbers to determine significance between the control arm and the treatment arms; however, we expect to collect useful information for future trials. It is assumed that equivalence will not likely be determined based on the sample size.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ambulatory
* Within 7 years post menopause
* Positive history of menopausal symptoms such as vasomotor symptoms or osteoporosis in a study subject unable to tolerate bisphosphonates
* FSH greater than 20 mIU/mL
* Intact uterus and at least one intact ovary
* Amenorrhea for 3 months or greater up to 7 years
* Normal pap smear results within 12 months
* Normal mammogram result within 12 months
* Agreeable to a 3 month washout period with no hormones prior to entering the trial
* Women who have no language barrier, are cooperative, and who can give informed consent before entering this study

Exclusion Criteria:

* Unwilling to take hormone replacement for the 12 month period
* Evidence of clinically significant psychiatric disorder by history/examination that would prevent the patient from completing the study.
* Active deep venous thrombosis, pulmonary embolism, or a history of these conditions
* Active or recent arterial thromboembolic disease
* Undiagnosed vaginal bleeding
* Hypersensitivity to ingredients in Prempro
* Patients with known current bone disorders other than primary osteoporosis
* Patients with pathological fractures
* Patients with suspected or history of carcinoma of the breast or estrogen dependent neoplasms such as endometrial carcinoma.
* Patients who have ≥ 5mm endometrial thickness by endovaginal (transvaginal) ultrasound.
* Patients who have impaired renal function evidenced by serum creatinine greater than 2.5 mg/dL.
* Patients who have impaired hepatic function evidenced by transaminase (AST/ALT) ≥2.5X upper limit
* Patients with severe malabsorption syndromes.
* Patients who consume an excess of alcohol or abuse drugs (an excess of alcohol is defined as more than four of any one or combination of the following per day: 30 mL distilled spirits, 340 mL beer, or 120 mL wine).
* Treatment with therapeutic doses of any of the following medications more recently than 3 months:

  * Estrogen
  * Calcitonin
  * Corticosteroids
  * Progestins
  * Progesterone
  * Lithium
  * Androgen
  * Heparin
  * Herbal menopause treatments
  * SERMS
  * Fluorides
  * Phosphate binding antacids
  * Bisphosphonates
  * Vitamin D 50,000IU
  * Anticonvulsants
* Patients who received any investigational drug within the proceeding month
* Tobacco use will not be allowed

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-02; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne A Drisko, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Limited sample size and high drop out rate make data obtained of marginal value. We will decide on a case by case review if data will be made available to requesting researchers. We recognize that data sharing includes protected health information and the deserved rights of individuals who participate in research. We will make every effort to protect these data at all times. Such data intended for broader use will be free of identifiers that would permit linkages to individuals, research participants or variables that could lead to deductive disclosure of the identify of individual subjects. This is in accordance for "Standards for Privacy of Individually Identifiable Health Information" - The Privacy Rule - HHS dated August 14, 2002. The Privacy Rule is a Federal regulation under the Health Insurance Portability and Accountability Act (HIPAA) of 1996 that governs the protection of individually identifiable health information.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Double blind single site pilot clinical trial conducted at academic medical center. Participants randomized to one of 4 arms by computer assignment conducted at independent site not enrolling subjects.
Pre-assignment Details: If participants were on hormone replacement at enrollment, needed to have 3 month washout period before randomization. Participants were required to be nonsmokers, have intact uterus, and be menopausal. Screening ultrasound of the uterus, bone density, screening metabolic panel, and baseline mammogram were required.
Groups:
- Participants Randomized to Arm 1: Participants in Arm 1 received Prempro, premarin .45mg, provera 1.5mg conjugated estrogens, medroxyprogesterone acetate Prempro, premarin, provera conjugated estrogens, medroxyprogesterone acetate: Prempro, premarin .45mg, provera 1.5mg conjugated estrogens, medroxyprogesterone acetate
- Participants Randomized to Arm 2: Participants in Arm 2 received compounded Estradiol .5mg, estriol 210mg, progesterone 100mg
  Estradiol , estriol , progesterone: Estradiol .5mg, estriol 210mg, progesterone 100mg
- Participants Randomized to Arm 3: Participants in Arm 3 received compounded estriol 2.5mg, progesterone 100mg
  estriol, progesterone: estriol 2.5mg, progesterone 100mg
- Participants Randomized to Arm 4: estradiol,progesterone
  estradiol,progesterone: estradiol,progesterone
Period: Overall Study
Arm/Group | Participants Randomized to Arm 1 | Participants Randomized to Arm 2 | Participants Randomized to Arm 3 | Participants Randomized to Arm 4
Started | 6 | 6 | 5 | 4
Completed | 2 | 1 | 2 | 4
Not Completed | 4 | 5 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — cancer unrelated to study discovered | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Arm 1: Prempro, premarin .45mg, provera 1.5mg conjugated estrogens, medroxyprogesterone acetate
  Prempro, premarin, provera conjugated estrogens, medroxyprogesterone acetate: Prempro, premarin .45mg, provera 1.5mg conjugated estrogens, medroxyprogesterone acetate
- Study Arm 2: Estradiol .5mg, estriol 210mg, progesterone 100mg
  Estradiol , estriol , progesterone: Estradiol .5mg, estriol 210mg, progesterone 100mg
- Study Arm 3: estriol 2.5mg, progesterone 100mg
  estriol, progesterone: estriol 2.5mg, progesterone 100mg
- Study Arm 4: estradiol,progesterone
  estradiol,progesterone: estradiol,progesterone
- Total: Total of all reporting groups
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 4 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 4 | 21
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 5 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Cholesterol
Description: To determine if bioidentical hormone replacement therapy is associated with change in lipid profiles (surrogate marker for cardiovascular disease) when compared to Prempro and provide safety data to proceed to larger trial. This was determined by evaluating lipid levels at baseline and during the 12-month treatment period. Participants' values were averaged at baseline and again at 12 months; the average of the baseline value was subtracted from the average at completion.
Time Frame: Baseline and month 12
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Study Arm 1: Menopausal women in first seven years of menopause randomized to arm 1 receive conjugated equine estrogens 0.45 mg combined with medroxyprogesteroneacetate 1.5 mg placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
- Study Arm 2: Menopausal women in first seven years of menopause randomized to arm 2 estradiol .5mg, estriol 2.0mg, progesterone 100mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
- Study Arm 3: Menopausal women in first seven years of menopause randomized to arm 3 estriol 2.5mg, progesterone 100mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
- Study Arm 4: Menopausal women in first seven years of menopause randomized to arm 4 estradiol 0.5 mg, progesterone 100 mg dosed orally / day placed in a placebo capsule to disguise contents from participant and study team. Drug dosed daily for 1 year. Screening FSH and PAP. Baseline mammogram, bone density, pelvic ultrasound, EKG, blood work for cholesterol panel (surrogate marker for cardiovascular disease), BUN/Creatinine. Repeated at 12 months. Safety check at 6 months includes BUN/creatinine, EKG, cholesterol panel, estradiol, progesterone levels.
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4
Number analyzed (Participants) | 2 | 1 | 2 | 4
mg/dL | 221.5 (12.5) | 221.5 (0) | 223 (26) | 165.5 (11)

2. Primary Outcome: Endometrial Measurement
Description: Baseline and 12 month follow up endovaginal ultrasound(completed at study site only) to evaluate endometrial stripe thickness for change on hormone therapy for all 4 arms. Endometrial thickness was measured in millimeters at baseline and again at 12 month completion. The average of the baseline value was subtracted from the average at completion for each group and reported in mm. Single participant in Arm 2: compared baseline to completion.
Time Frame: Baseline and month 12
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4
Number analyzed (Participants) | 2 | 1 | 2 | 4
mm | 13.0 (0) | 10.0 (0) | 2.5 (0.7) | 3.1 (0.7)

3. Primary Outcome: Number of Participants Without Change in Baseline and Follow up Mammograms
Description: Comparison at baseline and month 12 by descriptive analysis of breast mammograms. Assessing for changes in density and/or lesions for risk of breast stimulation from hormone replacement therapy. Mammogram readings for participants completing study in descriptive terms. Looking for significant change in breast tissue while on hormone therapy for 12 months. Those who had no change are counted below.
Time Frame: baseline and month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4
Number analyzed (Participants) | 2 | 1 | 2 | 4
Participants | 2 | 1 | 2 | 4

4. Secondary Outcome: Number of Participants Without Change in Baseline and Follow up Bone Density
Description: Comparison at baseline and month 12 by descriptive analysis of bone density. Assessing for changes in density related to hormone replacement therapy. Bone density readings for participants completing study in descriptive terms. Looking for significant change in bone density while on hormone therapy for 12 months. Those who had no change are counted below.
Time Frame: baseline and 12 months
Population: Only 7 participants completed both the baseline bone density and 12-month follow up bone density resulting in a discrepancy in evaluable numbers compared to other outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4
Number analyzed (Participants) | 1 | 1 | 2 | 3
Participants | 1 | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: Each participant had monitoring for adverse events from enrollment through the 1 year on trial.
Arm/Group | Study Arm 1 | Study Arm 2 | Study Arm 3 | Study Arm 4
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 2/5 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm 1 (N=6) | Study Arm 2 (N=6) | Study Arm 3 (N=5) | Study Arm 4 (N=4)
Abnormal vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes